CLINICAL TRIAL: NCT02915003
Title: A Partnership Approach to Enhance Health Care Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute for Health Care Reform (Unknown)
Responsible Party: Principal Investigator, Minal Patel, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00116683
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Insurance, Health
Keywords: health care navigation; health literacy; Affordable Care Act

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-health website intervention (Experimental): e-Health website embedded with short, culturally and locally-tailored videos informed by behavior change principles that will teach patients/families about: the importance and benefits of health insurance, ACA coverage provisions and local insurance options available to them, the specifics of the new law and how it affects them, and how to navigate local systems and resources to obtain and maintain health insurance.
  Interventions: Behavioral: E-health website
- Control (No Intervention): usual health insurance navigation, and ACA materials provided by social service agencies and clinics where individuals seek services.

INTERVENTIONS:
Behavioral: E-health website — e-Health website embedded with short, culturally and locally-tailored videos informed by behavior change principles that will teach patients/families about: the importance and benefits of health insurance, ACA coverage provisions and local insurance options available to them, the specifics of the new law and how it affects them, and how to navigate local systems and resources to obtain and maintain health insurance.
  Arms: E-health website intervention

SUMMARY:
With the help of local focus groups, the investigators are designing and testing a website to help urban people have better access to health care through understanding their insurance options better. They hypothesize that once individuals engage with the website and go through all of its modules, they will: 1) become more informed consumers of the ACA and its health insurance options; 2) enroll in an insurance plan; and 3) better leverage the benefits of their existing plans."

DETAILED DESCRIPTION:
The Affordable Care Act (ACA) has afforded millions of Americans with both greater access to and greater affordability of health insurance and its associated benefits. However, limited resources have been devoted for effective ACA outreach and enrollment - especially in states that did not create their own health insurance exchanges such as Michigan. Federally Qualified Health Centers (FQHCs) in Detroit are vital to meeting the health and medical care needs of the local community. However, they face long-term sustainability challenges, particularly related to their financial capacity, which can be augmented by increasing the number of insured patients that they serve.

The goal of the proposed project is to establish a new community-based participatory research (CBPR) partnership aimed at enhancing health care literacy of community residents of Detroit as it relates to the implementation of the ACA, through the design, implementation and evaluation of the effectiveness of an intervention trial. In accordance with the principles of CBPR, a Steering Committee will be established, involving four FQHCs and social service agencies working in Detroit, four community partner organizations, and academic members of the research team. The investigators will first conduct 9 focus groups with Detroit residents who use the local FQHCs and social service agencies and 1 focus group with health care navigators in order to inform the development of the e-Health intervention and better ascertain the healthcare literacy challenges residents face accessing information about the ACA. The investigators propose to develop and evaluate a healthcare literacy, e-Health intervention embedded with short, culturally and locally-tailored videos informed by behavior change principles that will teach patients/families about: the importance and benefits of health insurance, ACA coverage provisions and local insurance options available to them, the specifics of the new law and how it affects them, and how to navigate local systems and resources to obtain and maintain health insurance. They will recruit 240 patients/families seen at 4 local-area FQHC and social service sites to examine whether patient use of the website increases health care literacy and encourages individuals to enroll in health insurance plans. They will employ a randomized cross-over lagged research design where 120 patient/families seen at 2 FQHC and social service sites will be approached to use the website. The investigators will also identify 120 patients/families seen at 2 other sites who will serve as a lagged control group in the first segment of the study. Both the 120 intervention patients/families and the lagged control patient/families will be asked to complete a questionnaire about the ACA and other pertinent issues at the onset of the study. Six months later, they will again survey the patients in both groups (using the same survey instrument) to see whether any differences between the groups can be detected after 6 months. At that time, the 100 patient/families in the lagged control group will then be given the website (treatment) and they will follow them for 3 months. The investigators hypothesize that once individuals engage with the website and go through all of its modules, they will: 1) become more informed consumers of the ACA and its health insurance options; 2) enroll in an insurance plan; and 3) better leverage the benefits of their existing plans.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-64
2. identify as African American, Latino/Hispanic, or Arab American
3. access to a telephone

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline questionnaire measures of self-efficacy in navigating health insurance options at 6 and 9 months | baseline, 6 months, 9 months
  self-reported assessment of confidence in navigating several facets of health insurance that will be summed for a single score

SECONDARY OUTCOMES:
Change from baseline questionnaire measure of behavioral intention with health insurance navigation at 6 and 9 months | baseline, 6 months, 9 months
  participants will be asked if they intend to enroll in a health insurance plan or seek help at the time of assessment
Change from baseline measure questionnaire measure of Knowledge about the Affordable Care Act at 6 and 9 months | baseline, 6 months, 9 months
  participants will be asked a series of true/false statements about key provisions of the Affordable Care Act. A knowledge score will be generated based on the sum of responses from the knowledge questionnaire
Change from baseline use of questionnaire measures of beliefs around preventative health services use at 6 and 9 months | baseline, 6 months, 9 months
  participants will be asked if they have a usual source of care and have seen a doctor for routine care. Each item will be analyzed individually, and scores will be created for a sum of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Minal R Patel, PhD, MPH, Principal Investigator — University of Michigan